CLINICAL TRIAL: NCT07071870
Title: A Multicenter Prospective Randomized Controlled Non-Inferiority Trial Comparing Minimally Invasive SAIF Vertebral Reconstruction Technique Versus Spinal Fixation in Unstable Osteoporotic Vertebral Compression Fractures
Brief Title: RCT on the Efficacy and Safety of Minimally Invasive SAIF Technique vs Spinal Fixation in Unstable Osteoporotic Vertebral Fractures
Acronym: SAIF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eva Koetsier MD PhD (Other)
Collaborators: Prof. Dr. Med. Alessandro Cianfoni, MD PhD, Neurocenter of Southern Switzerland - Ente Ospedaliero Cantonale (EOC) (Unknown)
Responsible Party: Sponsor-Investigator, Eva Koetsier MD PhD, MD PhD LLM, Ospedale Regionale di Lugano
Organization: Ospedale Regionale di Lugano (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-02396
Record Dates: First submitted 2025-04-30; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Unstable Osteoporotic Vertebral Compression Fractures
Keywords: Stent-screw Assisted Internal Fixation (SAIF); Surgical stabilization

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stent-screw Assisted Internal Fixation (SAIF) (Experimental): SAIF technique, performed by percutaneous access, consists of, implanting vertebral body stents (VBS) under fluoroscopic guidance, followed by insertion of percutaneous, fenestrated, cement-augmented pedicular screws that act as anchors to the posterior elements for the cement/stent complex. The screws reduce the risk of stent mobilization in a non-intact vertebral body (VB) cortical shell and bridge middle column and pedicular fractures.
  Interventions: Procedure: Stent-screw Assisted Internal Fixation (SAIF)
- Surgical stabilization (Active Comparator): Spinal stabilization with augmented or non-augmented pedicle screws bridging the fractured vertebra, with or without (percutaneous) cement augmentation of the fractured vertebra, with or without reconstruction of the anterior column via anterior or lateral approach.
  Interventions: Procedure: Surgical stabilization

INTERVENTIONS:
Procedure: Stent-screw Assisted Internal Fixation (SAIF) — Implanting vertebral body stents (VBS), followed by insertion of percutaneous, fenestrated, cement-augmented pedicular screws
  Other Names: SAIF
  Arms: Stent-screw Assisted Internal Fixation (SAIF)
Procedure: Surgical stabilization — Spinal fixation with cement augmented pedicle screws bridging the fractured vertebra
  Arms: Surgical stabilization

SUMMARY:
Osteoporotic vertebral fractures (OVF) represent a significant cause of morbidity, mortality, decreased level of function and quality of life.

The most severe OVFs are unstable and in these cases surgical stabilization, with various techniques, is considered necessary to restore the physiological loading capacity of the spine, and allow fast and painless mobilization. Unfortunately, the elderly, osteoporotic patient population poses serious challenges to spinal surgery, due to tissue frailty and frequent comorbidities. The purpose of this study is to evaluate the effectiveness and safety of the SAIF intervention in comparison with multilevel surgical stabilization in participants with unstable OVFs.

DETAILED DESCRIPTION:
Osteoporosis is an increasing health problem worldwide with an enormous economic burden for society. Osteoporotic vertebral fractures (OVF) represent a significant cause of morbidity, mortality, decreased level of function and quality of life. Stable fractures with controllable pain can be managed conservatively, and only those that remain painful despite conservative treatment can be treated with minimally-invasive measures of vertebral augmentation (VA). At the other end of the spectrum, the most severe OVFs are unstable. In these cases standard vertebral augmentation techniques are generally considered an under-treatment and surgical stabilization, with various techniques, is considered necessary to restore the physiological loading capacity of the spine, and allow fast and painless mobilization. Unfortunately, this elderly, osteoporotic patient population poses serious challenges to spinal surgery, due to tissue frailty and frequent comorbidities. More specifically, all the surgical stabilization techniques include rigid posterior fixation of multiple spinal segments, but the reduced bone mechanical properties of osteoporotic patients can lead to hardware implant failure, new fractures, complications, and need of re-intervention.

On the other hand, treatment and reinforcement of the anterior spinal column, that should enhance posterior stabilization, requires a more invasive surgical approach, which carries a significant rate of complications and prolonged recovery times in this elderly population.

A recently described minimally-invasive interventional technique, called Stent-screw Assisted Internal Fixation (SAIF), can reconstruct, stabilize and restore axial load capability of the vertebral body affected by severe fractures, potentially obviating the need of a surgical multi-level rigid construct.

The study seeks primarily to determine whether the SAIF intervention is not inferior to surgical stabilization in improving quality of life in subjects with unstable OVFs at one year follow-up.

The principle secondary objective of this study is to evaluate whether the effect of the SAIF intervention on the radiological outcome is not inferior to surgical stabilization in subjects with OVFs.

Other secondary objectives are to compare both treatments in terms of safety, length of operation, blood loss, days of hospitalization postoperatively, pain, the intake of analgesics, disability and cost-effectiveness.

The total expected number of patients to randomized is 140, 70 per group. This ensures 80% power to test the hypothesis that SAIF is not inferior to surgical stabilization in increasing quality of life measured with the QUALEFFO questionnaire, assuming a standard deviation of 16 points, with a non-inferiority margin of 8 points. This also ensures over 90% power to exclude a non-inferiority margin of 4 degrees of kyphosis correction. The alpha for testing is set at 5%.

Estimated duration for the main investigational plan will be 60 months (from start of screening of first subject to last subject processed and finishing the study).

ELIGIBILITY:
Inclusion Criteria:

* one to two unstable OVFs* type OF 3-5** as assessed on CT scan, located between T2 and L5, of age <3 months or with persistent edema on STIR, or with pseudarthrosis, at the index level
* patients reporting pain upon mobilization
* a diagnosis of osteoporosis, based on a DEXA T-score ≤ -2.5, or on a spontaneous thoracolumbar vertebral fracture or a vertebral fracture caused by minor trauma
* able to read and speak the official language of the region of the site,
* informed consent

  * additional OVF without unstable features (OF 1-2) allowed ** OF-Classification

Exclusion Criteria:

* compressive neurologic symptoms such as myelopathy or radiculopathy with motor deficit
* acute infection
* spinal malignancy
* comorbid severe psychiatric conditions
* known or suspected non-compliance, drug or alcohol abuse
* known hypersensitivity or allergy to the investigational product
* inability to follow the procedures of the study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the Quality of Life questionnaire of the European Foundation of Osteoporosis (QUALEFFO) score. | at 12 months from baseline.
  The QUALEFFO score is patient-reported and comprises 41 items on five domains: pain, physical function, social function, general health perception, and mental function. All answers are standardized so that 1 represents the best and 5 (or 3, or 4) represents the worst quality of life.
  The total score is calculated by summing all answers of questions 1-41. The raw total score ranges from 41 to 205 and this is transformed to scores from 0 to 100. A high score indicates a poor quality of life.

SECONDARY OUTCOMES:
restoration of angular kyphosis at index level | pre-operative and at 1, 6 and 12 months follow up
  Restoration of angular kyphosis at index level (local kyphotic angle LKA and vertebral kyphotic angle VKA) comparing pre-operative with postoperative standing radiographs (local) and full spine standing radiographs at follow-up.
  This will be quantified as kyphosis correction at the index level in degrees. The non-inferiority margin is determined at 4 degrees.
vertebral body height restoration | Baseline and 1 day after the intervention
  Vertebral body height restoration (anterior VB, mid VB, post VB, or ratio of these) comparing pre- and post-operative computed tomography (CT) scan.
global kyphosis/lordosis | pre-operative and at 1, 6 and 12 months follow up
  Calculation of the Cobb angle at the thoracic and lumbar segments using a full spine stanting radiograph
Global Sagittal Balance | pre-operative and at 1, 6 and 12 months follow up
  Calculation of Sagittal Vertical Axis assessed with full spine stanting radiographs
length of operation | Perioperative
  minutes from skin insertion to skin closure during the tratment
blood loss | up to 1 week
  blood transfusion from the beginning of the intervention to discharge
days of hospitalization postoperatively | up to a week
  the number of days between the intervention and discharge. In case of outpatient (day surgery), the days of hospitalization are zero
back pain | at baseline and at 1, 3, 6 and 12 months follow up
  back pain measured with the numeric rating score (NRS): 11-point NRS ranging from 0 (no pain at all) to 10 (the worst imaginable pain). A score of zero (0) will indicate that the patient is pain free, while a score of ten (10) will indicate that they are experiencing the worst pain imaginable.
the intake of analgesics using the Medication Quantification Scale (MQS). | at baseline and at 1, 3, 6 and 12 months follow up
  The score is calculated for each medication by taking a consensus-based detriment weight for a given pharmacologic class and multiplying it by a score for dosage. The calculated values for each medication are then summed for a total MQS score
disability using Roland-Morris disability questionnaire (RMDQ) | at 1, 3, 6 and 12 months follow up
  24 items that assess functional status over the past 24 hours in patients with back pain.
  The total score ranges from 0 to 24:
  0 = no disability 24 = maximum disability related to low back pain. A change in 2-3 points on the RDQ is considered the minimum clinically important change.
cost-effectiveness | up to 12 months.
  two outcomes are combined: the quality-adjusted life year (QALY) that takes into account the quantity (longevity/mortality) and the health-related quality of life (HRQoL), and costs that include health care related costs, costs to patients and family, and costs related to paid and unpaid home care.

OTHER OUTCOMES:
Safety outcomes | up to 12 months.
  adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- EOC Lugano, Lugano, Canton Ticino, Switzerland